CLINICAL TRIAL: NCT04510636
Title: Phase 2 Study Evaluating the Safety and Efficacy of Pembrolizumab (KEytruda) in Combination With Bendamustine (TREanda) in Relapsed/Refractory Hodgkin Lymphoma
Brief Title: Study of Pembrolizumab With Bendamustine in Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KEsTREL-01; CAPCR 20-5231 (Other: University Health Network)
Record Dates: First submitted 2020-08-09; First posted 2020-08-12 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Classical Hodgkin Lymphoma; Relapsed Cancer; Refractory Cancer
MeSH Terms: conditions — Recurrence; Neoplasms | interventions — pembrolizumab; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab and Bendamustine (Experimental): The study drugs will be given in 3 week periods called cycles.
  Pembrolizumab is available in powder form or as a liquid for infusion. Pembrolizumab at a dose of 200 mg will be given over 30 minutes, once every cycle for up to 35 cycles (approximately 24 months).
  Bendamustine is available in powder form for injection. Bendamustine at a dose of 90 mg/m2 will be given over 60 minutes, on Days 1 and 2 of every cycle for up to 6 cycles.
  Interventions: Drug: Pembrolizumab; Drug: Bendamustine Hydrochloride

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab is a intravenously administered humanized monoclonal antibody that blocks the interaction between PD-1 and its ligands, PD-L1 and PD-L2.
  Other Names: KEYTRUDA
Drug: Bendamustine Hydrochloride — Bendamustine is a unique alkylating agent with substantial activity in hematologic malignancies.
  Other Names: TREANDA

SUMMARY:
This is a phase 2 open-label study to test the safety and effectiveness of combining pembrolizumab and bendamustine in patients with relapsed (cancer that has come back or started getting worse) or refractory (cancer that is not responding or has stopped responding to treatment) Hodgkin lymphoma.

DETAILED DESCRIPTION:
Pembrolizumab and bendamustine will be explored as a safe and effective treatment for these patients.

Although current treatment options are available for patients in the relapsed state, once these therapies fail or are not tolerated, treatment options are quite limited.

Pembrolizumab and bendamustine have both shown activity when used as a single agent as treatment for Hodgkin Lymphoma. Their side effect profiles also do not overlap, which makes them ideal to combine, with an intent to increase the amount and duration of complete responses while limiting the toxicities experienced by patients.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial and adhere to trial procedures.
* Have histologically confirmed relapsed (disease progression after most recent therapy) or refractory (failure to achieve complete response [CR] or partial response [PR] to most recent therapy) classical Hodgkin Lymphoma).
* Must have received at least standard first line chemotherapy for classical Hodgkin Lymphoma, containing an anthracycline.
* Must have failed or declined autologous stem cell transplantation (ASCT), or not be a candidate for ASCT.
* May have received prior therapy with pembrolizumab (or an equivalent checkpoint inhibitor or anti-PD-L1 antibody), but not in combination with bendamustine.
* May have received a prior autologous stem cell transplant but must be at least ≥100 days post-auto-transplant, and all transplant- related adverse events must have resolved to a grade 1 or less, and patients are not on immunosuppression, and meet all other eligibility criteria.
* Must have measurable or evaluable disease.
* Must have Eastern Cooperative Group (ECOG) performance status 0-1.
* Must have an estimated life expectancy of greater than 90 days.
* Demonstrate adequate organ and bone marrow function.
* If female of child-bearing potential, must have a negative pregnancy test within 72 hours prior to the first dose of study treatment.
* All participants must be willing to use adequate contraception for the duration of treatment with study drugs and continue for 120 days after the last dose of study drug.
* Must be available for treatment, assessment and follow-up.

Exclusion Criteria:

* There is known severe (≥ Grade 3) hypersensitivity to pembrolizumab or bendamustine.
* Patient receiving any other investigational agents, or has participated in a study of an investigational agent and has received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Patient is receiving any other, non-investigational, chemotherapy, radiotherapy, small molecule, or biologic agent within 4 weeks of the first dose of treatment, or who has not recovered from adverse events due to a previously administered agent.
* Patient has had a prior monoclonal antibody within 4 weeks prior to first dose of therapy in the study, or who has not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Patient has received pembrolizumab, or another anti-PD1, or anti-PD-L1, anti-PD-L2, anti-CD137, anti-CTLA-4, or anti-OX-40 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways, with disease progression whilst on therapy, or within 3 months of completion of this line of therapy, without intervening systemic therapy (including chemotherapy, antibody drug conjugates or other targeted agents).
* Patient has received prior treatment with bendamustine, either as monotherapy or as part of a combination regimen.
* Patient has undergone prior allogeneic hematopoietic stem cell transplant.
* Patient has another concurrent active malignancy (excluding non-melanoma skin cancer or carcinoma in situ of the cervix that has undergone potentially curative therapy), and must be disease-free and off treatment for > 3 years.
* Patient has known active central nervous system or meningeal disease.
* Patients with active or past documented autoimmune disease that has required treatment in the past 2 years.
* Patient is receiving systemic steroid therapy at a dose of > 10 mg/day of prednisone (or equivalent) for 7 days prior to day 1 of study treatment.
* Has an uncontrolled co-existing illness, including but not limited to: ongoing or active infection requiring systemic therapy; systemic congestive heart failure Class III or IV by NYHA criteria; unstable angina pectoris or cardiac arrhythmia; in patients status post allogeneic transplantation uncontrolled GVHD.
* Patient has a history of (non-infectious) pneumonitis that has required steroid treatment, or concurrent active pneumonitis.
* Patient is pregnant, or nursing, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of pembrolizumab and/or bendamustine.
* Has a known history of Human Immunodeficiency Virus (HIV), active tuberculosis (TB, Mycobacterium tuberculosis), or active hepatitis B or hepatitis C.
* Patient has received a live vaccine within 30 days prior to first dose of study drugs.
* Patient is eligible for autologous or allogeneic stem cell transplant, unless patient has declined this, therefore rendering themselves ineligible for stem cell transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2021-12-20 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 5 years
  Complete response + partial response
Complete response rate as determined by Lugano criteria | 5 years
  Assessed by positron emission tomography (PET)/computed tomography (CT) scans

SECONDARY OUTCOMES:
Incidence of adverse events | 5 years
  duration from start of study until end
Overall survival rate | 5 years
  for the duration of study
Progression-free survival rate | 5 years
  for the duration of study
Average duration of response | 5 years
  for the duration of study

CONTACTS AND LOCATIONS:
Overall Officials: John Kuruvilla, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No